CLINICAL TRIAL: NCT01171729
Title: A Phase I/IIa Study of Autologous Cell-based Vaccine Therapy With CreaVax-PC in Hormone-Refractory Metastatic Prostate Cancer Patients With PSA Relapse to Evaluate the Safety and Efficacy
Brief Title: Autologous Dendritic Cell Therapy for Hormone-Refractory Metastatic Prostate Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Collaborators: National Cancer Center, Korea (Other Government)
Responsible Party: Chul Won Jung, MD, Samsung Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006-10-030
Record Dates: First submitted 2010-07-27; First posted 2010-07-28 (Estimated); Last update posted 2010-08-11 (Estimated); Status verified 2010-07

CONDITIONS: Prostatic Cancer
Keywords: Prostate cancer; PSA; Hormone refractory prostatic cancer
MeSH Terms: conditions — Prostatic Neoplasms; Prostatic Neoplasms, Castration-Resistant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: Autologous dendritic cell — Autologous dendritic cells pulsed with prostate cancer antigen and KLH
  Other Names: CreaVax-PC

SUMMARY:
This is an open label, Phase I/IIa trial of immunotherapy with CreaVax-PC as treatment in men with hormone-Refractory Metastatic Prostate Cancer.

DETAILED DESCRIPTION:
CreaVax-PC consisted of antigen (PSA, PAP and KLH) primed dendritic cell is an investigational product designed to activate a man's immune response, so they can detect prostate cancer cells and initiate an immune response against prostate cancer antigens.

If patients decide to participate and are eligible, they will be enrolled in the study and will receive active product (CreaVax-PC). In detail, patients will receive CreaVax-PC injection at intervals of 3 weeks, maximum 6 times during 21 weeks. PSA increase rate is a primary evaluation variables and tumor suppression effect is secondary evaluation variables. We also evaluate time to progression, overall survival and immune response.

ELIGIBILITY:
Inclusion Criteria:

* 1) Histological confirmed prostatic carcinoma patient
* 2) Hormone non-respondence ex1) Although treatment PSA ≥ 5ng/ml ex2) PSA level were measured two times ex3) Prior one year radiology were processed
* 3) Just 18 years over
* 4) Has a score ≤1 on the ECOG Performance Scale
* 5) Expected survival life time ≥ 6month
* 6) Adequate bone marrow function hemoglobin ≥ 10.0g/dL , leukocyte count ≥ 4,000/mm3 thrombocyte ≥ 100,000/mm3
* 7) Adequate blood coagulation function PT(INR) < 1.5, aPTT< 1.5 x control
* 8) Adequate kidney function Normal blood upper level Creatinine ≤ 1.5 times
* 9) Adequate liver function Normal blood upper level AST/ALT ≤ 1.5 times
* 10) Autoimmune antibody system don't have disorder ex) anti-nuclear antibody, anti-thyroglobulin antibody negativity
* 11) Person who didn't treat prior 6 weeks operation, radiotherapy treatment,immunotherapy or chemotherapy
* 12) Patient who voluntarily participated clinical trial and confirmed a written consent

Exclusion Criteria:

* 1) Having other malignancy or previous history of malignancy
* 2) Brain metastases patient
* 3) Having autoimmune disease or its history
* 4) Pyrexia, rigor, leukocytosis infectious disease
* 5) HBsAg, anti-HCV, HIV positive patient
* 6) Myocardial infarction, cardiac insufficiency, other severe heart disease and non-controlled hypertension
* 7) Severe and active medical disease
* 8) Mental history disease or epilepsy
* 9) Patients participated other clinical trial within 4 weeks
* 10) Patients impossible to participate this trial by investigator's decision
* 11) Patients who received immunosuppressant such as steroid, cyclosporin A, azathioprine within 6 weeks

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2006-07; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
PSA increment and absolute PSA response | 12 weeks
  PSA response evaluation at 12 weeks and follow up response evaluation at 21 weeks

SECONDARY OUTCOMES:
Time to Progression | DC Injection to time to progression or death
Overall Survival | Patients will be followed until death
Immune Response(DTH response, Interferon-gamma Elispot assay, proliferation assay, ELISA) | weeks 0, 12, 21
Clinical response | week 0, 12, 21
  Clinical course of participants as measured by bone scans and CT

CONTACTS AND LOCATIONS:
Overall Officials: J C W, M.D,Ph.D, Principal Investigator — Samsung Medical Center
Locations (2):
- South Korea (2):
  - National Cancer Center, Gyeonggi-do, 323 Ilsan-ro Ilsandong-gu Goyang-si
  - Samsung Medical Center, Seoul, Gangnam-Gu, Ilwon-Dong